CLINICAL TRIAL: NCT00775840
Title: Candesartan "Added" Therapy for Treatment Optimization of Symptomatic Heart Failure With Diastolic Dysfunction in Diabetic and Hypertensive Patients A Randomized, Placebo-controlled, Double-blind, Parallel-group and Multicenter Clinical Phase III Study Investigating the Effects on NT-proBNP Over 6 Months
Brief Title: Efficacy of Candesartan on Symptomatic Heart Failure in Treating Diabetic and Hypertensive Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma Gmbh, Aachen (Germany)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLO K026; 2007-003070-26 (EudraCT Number); D-CAN-546 (Other: Takeda ID); U1111-1113-9515 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Heart Failure
Keywords: Cardiac Failure; Congestive Heart Failure; Drug Therapy; Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Heart Failure; Hypertension; Diabetes Mellitus | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candesartan QD + Heart Failure Therapy (Experimental): (with angiotensin-converting enzyme-inhibitors/beta-blockers)
  Interventions: Drug: Candesartan
- Placebo QD + Heart Failure Therapy (Placebo Comparator): (with angiotensin-converting enzyme-inhibitors/beta-blockers)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candesartan — Candesartan up to 32 mg, tablets, orally, once daily and ongoing angiotensin-converting enzyme inhibitor/beta-blocker therapy for up to 24 weeks.
  Other Names: BLOPRESS®
  Arms: Candesartan QD + Heart Failure Therapy
Drug: Placebo — Candesartan matching-placebo tablets, orally, once daily and ongoing angiotensin-converting enzyme inhibitor/beta-blocker therapy for up to 24 weeks.
  Arms: Placebo QD + Heart Failure Therapy

SUMMARY:
The purpose of this study is to determine the effects of candesartan, once daily (QD), on the N-terminal pro-B-type Natriuretic Peptide laboratory marker in subjects with symptomatic heart failure with diastolic dysfunction.

DETAILED DESCRIPTION:
Heart diseases are the number one cause of death in developed countries and in particular chronic or congestive heart failure is the leading cause of hospitalization in patients older than 65 years. It is still increasing in prevalence and, in spite of significant advances in therapy, mortality rates remain high: 30% to 40% of patients with advanced disease, and 5% to 10% of patients with mild symptoms will die within 5 to 10 years.

A relevant proportion of the heart failure patients (30 - 50%) suffering from edema and dyspnea have normal or minimally impaired left ventricular ejection fraction (preserved left ventricular ejection fraction) with diastolic abnormalities in echocardiography. Features of diastolic dysfunction are the stiffness, the decreased compliance and the impaired relaxation of the left ventricle. As a result, the left ventricle has a limited filling capacity during a normal left atrial pressure.

Hypertension and/or diabetes are the most predisposing conditions whereas left ventricular hypertrophy is regarded as the linking intermediate pathological condition. Moreover, recent studies showed that patients with symptomatic heart failure and an ejection fraction greater than 40% have a poor prognosis with relatively high mortality and hospitalization rates. Thus, in hypertensive patients, diastolic dysfunction has shown to be a predictor of morbidity.

Diastolic dysfunction is also a frequent finding in type 2 diabetes without symptoms and signs of heart disease. As long as it is independent of ischemic heart disease, it is presumably due to diabetic cardiomyopathy. Once aggravated to heart failure, diastolic dysfunction often coexists with systolic dysfunction as a consequence of coronary artery disease with a limited coronary reserve.

This study will determine whether pharmacological intervention into the Renin Angiotensin Aldosterone System exerted by the Angiotensin-Receptor Blocker Candesartan on top of an Angiotensin-Converting Enzyme Inhibitor-based therapy may lead to a significant drop of N-terminal pro-B-type Natriuretic Peptide. This neurohormonal laboratory marker is sufficient enough to simultaneously indicate the improvement of the causing diastolic dysfunction and associated heart failure symptoms as assessed by objective echocardiographic and clinical parameters.

Total time for participants in this study is approximately 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2 - insulin dependent or orally treated or managed by diet for at least 3 Months.
* Normotension or controlled hypertension with sitting Systolic Blood Pressure less than 140 mmHg and/or sitting Diastolic Blood Pressure less than 90 mmHg.
* Regular sinus rhythm or atrial fibrillation with a medicamental-achieved rate control of less than 100 bpm as confirmed by electrocardiogram recordings.
* Echocardiographic evidence of a preserved Left Ventricular Ejection Fraction greater than or equal to 45% (assessed by the modified Simpson method), with further doppler-echocardiographic criteria for diastolic dysfunction grade I-IV.
* New York Heart Association classification of II or III in a stable condition since at least 3 months.
* Existing background heart failure therapy with an Angiotensin-Converting Enzyme Inhibitor alone or together with further preparations in a constant regimen since at least 1 month, in case of beta-blockers since at least 3 months.
* N-terminal pro-B-type Natriuretic Peptide greater than or equal to 250 pg/ml measured at screening visit or collected from a dated previous laboratory document not older than 3 months.
* No previous therapy with Angiotensin-Receptor Blockers during the last 4 weeks prior to the study.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Impaired renal function (serum creatinine greater than 2.2 mg/dl or greater than 194 μmol/l).
* Known bilateral renal artery stenosis or interventional treatment for renal artery stenosis in the last year.
* State after kidney transplantation.
* Serum potassium greater than 5.5 mmol/l or glycosylated hemoglobin greater than 9.5 %.
* Cor pulmonale or primary pulmonary disease with dyspnea at rest.
* Known disposition to episodes of symptomatic hypotension or sitting Systolic Blood Pressure less than 95 mmHg at baseline.
* Acute coronary syndrome or any form of unstable chronic Coronary Artery Disease where the indication of a coronary intervention is either planned in short or medium term or can not be clearly excluded for the period of the study.
* Any history of: myocardial infarction, previous Percutaneous Transluminal Coronary Angioplasty with revascularization, stent implantation, Coronary Artery Bypass Graft or open heart surgery.
* Tachycardia at rest greater than 100 bpm as confirmed by electrocardiogram recordings.
* Known clinically relevant rhythm disorders (e.g., tachyarrhythmias, salves of supraventricular or ventricular extrasystoles or atrial fibrillation without ventricular rate control) or symptoms suggesting a significant rhythm disorder (e.g., recurrent syncopes).
* Primary valvular diseases and/or restrictive or obstructive cardiomyopathy.
* Existing ventricular assist devices.
* Relevant liver diseases (cholestasis or alanine aminotransferase/aspartate aminotransferase greater than 2 times the upper limit of normal or gamma- glutamyltransferase greater than 3 times the upper limit of normal).
* History of primary hyperaldosteronism, of cancer in the last 5 years or of another wasting disease with life expectancy of less than 2 years.
* Known hypersensitivity to Candesartan Cilexetil.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Need for maintenance therapy with Non-steroidal anti-inflammatory drugs or Cox-2-inhibitors.
  * Use of other Angiotensin-Receptor Blockers.
* Any history of life-threatening diseases.
* History of drug addiction and/or an extensive use of alcohol.
* Acute coronary syndrome or unstable angina pectoris and any coronary artery disease that was not stable during the last 3 months prior to inclusion.
* Patients who are dependent on a permanently paced pacemaker (i.e. a patient with a device that is not pacing during the echocardiographic examination can enter the study).
* Open heart surgery for other reasons than coronary revascularization
* Participation in another clinical investigation within 30 days prior to enrolment or for the course of the present study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The change from Baseline in N-terminal pro-B-type Natriuretic Peptide biomarker. | Week 24 or Final Visit.

SECONDARY OUTCOMES:
Mean change in N-terminal pro-B-type Natriuretic Peptide (log-transformed). | Weeks 6 and 24 or Final Visit.
Change from Baseline in Short Form-36 Health Survey score. | Week 24 or Final Visit.
Change from Baseline in Cystatin C. | Week 24 or Final Visit.
Change from Baseline in Adiponectin. | Week 24 or Final Visit.
Change from Baseline in Glycosylated Hemoglobin. | Week 24 or Final Visit.
Change from Baseline in Urinary Albumin Excretion. | Week 24 or Final Visit.
Change from Baseline in estimated Glomerular Filtration Rate and Cystatin C. | Week 24 or Final Visit.
Mean Change in New York Heart Association classification results. | Week 24 or Final Visit.
Body Weight. | Week 24 or Final Visit.
Blood Pressure. | Week 24 or Final Visit.
Echocardiograms. | Week 24 or Final Visit.
Correlations of N-terminal pro-B-type Natriuretic Peptide with New York Heart Association Classification Results. | Week 24 or Final Visit.
Correlations of N-terminal pro-B-type Natriuretic Peptide with short Form-36 Health Survey Score. | Week 24 or Final Visit.
Correlations of N-terminal pro-B-type Natriuretic Peptide with Blood Pressure Results. | Week 24 or Final Visit.
Subgroup evaluations regarding beta-blocker therapy and New York Heart Association class (II/III). | Week 24 or Final Visit.
Subgroup evaluations in terms of the different possible dosages of study medication. | Weeks 6 to 24 or Final Visit.
Subgroup evaluations based on different baseline levels of estimated Glomerular Filtration Rate. | Week 24 or Final Visit.
Subgroup evaluations based on different baseline levels of Cystatin C. | Week 24 or Final Visit.
Subgroup evaluations based on different baseline levels of N-terminal pro-B-type Natriuretic Peptide. | Week 24 or Final Visit.
Comparison from Baseline on the concomitant use of Loop Diuretics. | Weeks 6 and 24 or Final Visit.
Transition from sinus rhythm to permanent atrial fibrillation based on electrocardiogram recordings. | Week 24 or Final Visit.
Progression of preserved (Left Ventricular Ejection Fraction greater than or equal to 45%) to impaired systolic dysfunction (Left Ventricular Ejection Fraction less than 45%), based on echocardiographic results. | Week 24 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Pharma Gmbh, Aachen (Germany)
Locations (37):
- Germany (37):
  - Bad Friedrichshall, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Ludwigsburg, Baden-Wurttemberg
  - Bad Homburg, Hesse
  - Bad Nauheim, Hesse
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Giessen, Hesse
  - Kassel, Hesse
  - Limburg an der Lahn, Hesse
  - Melsungen, Hesse
  - Mühlheim am Main, Hesse
  - Wiesbaden, Hesse
  - Nienburg, Lower Saxony
  - Northeim, Lower Saxony
  - Weyhe, Lower Saxony
  - Essen, North Rhine-Westphalia
  - Gelsenkirchen, North Rhine-Westphalia
  - Gladbeck, North Rhine-Westphalia
  - Langenfeld, North Rhine-Westphalia
  - Paderborn, North Rhine-Westphalia
  - Siegen, North Rhine-Westphalia
  - Bad Kreuznach, Rhineland-Palatinate
  - Neukirchen, Saarland
  - Dresden, Saxony
  - Hartmannsdorf, Saxony
  - Leipzig, Saxony
  - Leisnig, Saxony
  - Machem, Saxony
  - Markkleeberg, Saxony
  - Riesa, Saxony
  - Wermsdorf, Saxony
  - Coswig, Saxony-Anhalt
  - Berlin, State of Berlin
  - Erfurt, Thuringia
  - Jena, Thuringia
  - Nordhausen, Thuringia